CLINICAL TRIAL: NCT00523965
Title: A Randomised, Open-label, Parallel-group, Safety and Efficacy Study to Evaluate Different Combination Treatment Regimens (Co-administration), of AmBisome, Paromomycin and Miltefosine in Visceral Leishmaniasis (VL)
Brief Title: Combination Therapy in Indian Visceral Leishmaniasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Banaras Hindu University (Other)
Collaborators: Drugs for Neglected Diseases (Other); Rajendra Memorial Research Institute of Medical Sciences (Other)
Responsible Party: Shyam Sundar, Drugs for Neglected Diseases Initiative
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VLCombo 07
Record Dates: First submitted 2007-08-31; First posted 2007-09-03 (Estimated); Last update posted 2010-05-26 (Estimated); Status verified 2009-01

CONDITIONS: Leishmaniasis, Visceral
Keywords: Kala-azar; miltefosine; liposomal amphotericin B
MeSH Terms: conditions — Leishmaniasis, Visceral | interventions — amphotericin B, deoxycholate drug combination; liposomal amphotericin B; miltefosine; Paromomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A (Experimental): AmBisome 5 mg/kg iv infusion over 2 h x 1 day (single dose) + oral miltefosine 50mg once daily (< 25 kg body weight) or twice daily ( > 25 kg body weight) or 2.5 mg/kg for children under 12 years, for 7 days on day 2-8
  Interventions: Drug: Liposomal Amphotericin B with Miltefosine
- B (Experimental): AmBisome 5mg/kg iv infusion over 2 h x 1 day (single dose) + paromomycin sulfate 15 mg/kg/day i.m for 10 days, on day 2-11
  Interventions: Drug: Liposomal Amphotericin B and Paromomycin Sulfate
- C (Experimental): oral miltefosine 50mg once daily (< 25 kg body weight) or twice daily ( > 25 kg body weight) or 2.5 mg/kg for children under 12 years, for 10 days + Paromomycin sulfate 15 mg/kg/day im. for 10 days
  Interventions: Drug: miltefosine + Paromomycin sulfate
- D (Active Comparator): amphotericin B deoxycholate at 1 mg/kg every other day for 15 infusions
  Interventions: Drug: amphotericin B deoxycholate

INTERVENTIONS:
Drug: amphotericin B deoxycholate — Amphotericin B deoxycholate 1 mg/kg on alternate days for 15 infusions
  Arms: D
Drug: Liposomal Amphotericin B with Miltefosine — Liposomal Amphotericin B 5 mg Miltefosine 50 mg twice daily if patient weighs equal to or > 25 kg Miltefosine 50 mg once daily if patient weighs <25 mg
  Arms: A
Drug: Liposomal Amphotericin B and Paromomycin Sulfate — AmBisome 5mg/kg iv infusion over 2 h x 1 day (single dose) + paromomycin sulfate 15 mg/kg/day i.m for 10 days, on day 2-11
  Arms: B
Drug: miltefosine + Paromomycin sulfate — oral miltefosine 50mg once daily (< 25 kg body weight) or twice daily ( > 25 kg body weight) or 2.5 mg/kg for children under 12 years, for 10 days + Paromomycin sulfate 15 mg/kg/day im. for 10 days
  Arms: C

SUMMARY:
Rationale

The overall objective of this trial is to identify a safe and effective combination, (co-administration) short course treatment for the treatment of VL which could be easily deployed in a control programme. The hypothesis is that the combination treatment is as effective or better than the 5 mg/kg single dose of AmBisome and will reduce the risk of parasite resistance occurring. Safety and tolerability should be such that the combination can be easily deployed.

Objective

The specific primary and secondary objectives are as follows:

Primary objective:

To identify a short course combination treatment regimen which is at least as effective as a single dose of AmBisome 5mg/kg

Secondary objective:

To compare safety and tolerability of the various treatments measured by vital signs, blood biochemistry, (renal and liver function tests) haematology, spontaneous and elicited adverse event reporting

Primary Endpoint:

The primary efficacy endpoint variable is parasitological clearance 2 weeks after start of treatment with no relapse during follow up and no clinical signs or symptoms of VL at 6 months post treatment.

Parasitology is only carried out at any time during follow-up or at six months post treatment if there are signs or symptoms of VL infection.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 5 years old with symptoms and signs of kala-azar (fever, weight loss, splenomegaly) and parasites demonstrated by microscopy in splenic aspirate smear

Exclusion Criteria:

* Pregnant or breast-feeding women
* Individuals seropositive to HIV or individuals with a serious concurrent infection such as tuberculosis or bacterial pneumonia.
* Women of child-bearing age will be counseled about adequate birth control during and for three months after miltefosine treatment and provided with a satisfactory method of contra-ception.
* Granulocyte count < 1,000/mm3, hemoglobin < 5 g/dL or platelet count < 40,000/mm3
* Hepatic transaminases or total bilirubin greater than three times normal
* Serum creatinine > 2.0 mg/dL
* Prothrombin time > 5 seconds above control
* Inability of subject or guardian to provide written informed consent

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 624 (Estimated)
Dates: Start 2007-09; Primary Completion 2009-08 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Final cure at six month follow up | 18 months
Cure at six month follow up | 12 months

SECONDARY OUTCOMES:
Initial cure at the end of treatment | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Shyam Sundar, MD, Principal Investigator — Institute of Medical Sciences, Banaras HIndu University; P K Sinha, MD, Principal Investigator — Rajendra Memorial Research Insititute of Medical Sciences
Locations (1):
- Kala-azar Medical Research Center, Muzaffarpur, Bihar, India